CLINICAL TRIAL: NCT04812704
Title: Suppléments protéinés en Association d'un Programme de préhabilitation Avant la Prise en Charge Chirurgicale d'un Cancer
Brief Title: Protein Supplements in Association With Prehabilitation Program for Cancer Patients Before Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion difficulty
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Deswysen Yannick, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/19JAN/022
Record Dates: First submitted 2021-03-05; First posted 2021-03-24 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Cancer; Surgery; Prehabilitation
MeSH Terms: conditions — Neoplasms | interventions — Whey Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional complement (Experimental): A prospective study will be carried out including adult patients with neoplasia who should benefit in their therapeutic strategy from oncological surgery. About fifty patients will be recruited in the oncology / surgery department at the Saint-Luc University Clinics in Brussels. Patients will be assessed at the initial consultation and after the pre-habilitation period, ie the day before the operation.
  Dietary monitoring will be carried out in parallel with a physical and respiratory preparation program (prehabilitation) and the intake of protein nutritional supplements in the form of powder to be diluted will be carried out after each exercise session.
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Whey protein — Patient receive protein supplement in liquid form after each exercice session

SUMMARY:
The aim of study is to analyse the feasibility of the use of nutritionnal complements after exercices before surgery for cancer.

Body composition, muscle function and muscle mass will be analyse too.

DETAILED DESCRIPTION:
A prospective study will be carried out including adult patients with neoplasia who should benefit in their therapeutic strategy from oncological surgery. About fifty patients will be recruited in the oncology / surgery department at the Saint-Luc University Clinics in Brussels. Patients will be assessed at the initial consultation and after the pre-habilitation period, ie the day before the operation.

Dietary monitoring will be carried out in parallel with a physical and respiratory preparation program (prehabilitation) and the intake of protein nutritional supplements in the form of powder to be diluted will be carried out after each exercise session.

ELIGIBILITY:
Inclusion Criteria:

* patient with operable cancer
* patient inform consent
* min 18 years old
* french or english speaking

Exclusion Criteria:

* neuromuscular pathology
* cardiorespiratory or orthopedic pathology that prevents physical activity
* cognitive or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Adhesion rate of the use of nutritionnel complements after exercices before surgery for cancer | 3 weeks
  The feasibility of this outcome will be assess by the adhesion rate : (number of protein shots taken) / (number of protein shots prescribed). The adhesion will be validated if> 75% of the holds are respected.

SECONDARY OUTCOMES:
Body composition (lean and fat mass) | Once at the inclusion and once the day before surgery (3 weeks)
  Evaluated by an impedancemetry balance : pourcentage of lean and fat mass
Muscle function | Once at the inclusion and once the day before surgery (3 weeks)
  This variable will be studied by the 6-minutes walk test (meters)
Nutritional biological markers | Once at the inclusion
  These variables will be studied by: prealbumin (g/L) and albumin (g/L) measures
Antropometric markers - height | Once at the inclusion and once the day before surgery (3 weeks)
  Height (meters)
Muscle strength | Once at the inclusion and once the day before surgery (3 weeks)
  This variable will be studied by the hand grip test (kilograms)
Antropometric markers - weight | Once at the inclusion and once the day before surgery (3 weeks)
  Weight (kilograms)
Antropometric markers - BMI | Once at the inclusion and once the day before surgery (3 weeks)
  BMI (kg/m²) :weight and height will be combined to report BMI in kg/m²

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Deswysen, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No